CLINICAL TRIAL: NCT05324020
Title: Improving Oral Hormonal Therapy Adherence in Breast Cancer Survivors by Using eHealth as a New Intervention Tool
Brief Title: eHealth Intervention for Medication Adherence in Breast Cancer Survivors
Acronym: Edherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Centre Hospitalier du Luxembourg (Other); Centre Hospitalier Emile Mayrisch (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CNER 202107/05
Record Dates: First submitted 2022-02-23; First posted 2022-04-12 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Patient-physician communication; cancer survivor; eHealth; telemedicine; digital health; medication adherence; medication compliance
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E- Health medication adherence Intervention group (Experimental): 3 Month monitoring adherence and side-effect management using an eHealth intervention . Participants are in contact with there clinical care team which intervene in cases of non-adherence and/or side-effect reporting.
  Interventions: Behavioral: Medication adherence eHealth intervention

INTERVENTIONS:
Behavioral: Medication adherence eHealth intervention — The eHealth intervention consists a Medication Event Monitoring Systems (MEMS®) Helping Hand and MEMS Adherence Software application. The eHealth intervention will support BCS to adhere to their OHT (i) by alerting them to take their OHT, and (ii) by allowing patient-physician communication.
  The eHealth intervention comprises a questionnaire that should be filled-out weekly and that informs about the presence and severity of side effects. These data are collected in real-time and monitored on a weekly basis by the clinical research nurse (CRN) in charge of the study. In case of an alert, meaning recurrent non-adherence and/or reporting of side-effects, the CRN will contact the breast cancer nurse (BCN) in charge of the patient. Thus the BCN will contact the patient by phone to check on their health status and together define the future procedures (behavioral strategies).

SUMMARY:
Tamoxifen and aromatase inhibitors are two oral hormonal therapies (OHT) that decrease the risk of breast cancer recurrence by over 30 %. Their efficacy however strongly depends on the duration of use (5 to 10 years). Earlier work demonstrated that the longer an individual is not taking her OHT the less likely she is to restart her therapy.

Thus, identifying the moment of treatment interruption in real-time and being able to contact the patient at these specific time-points may be the key to effective health interventions by improving medication adherence to reduce BC recurrence - therefore, increasing overall Breast Cancer survival (BCS). EHealth technologies may be a very effective mean to identify these interruptions in a real-time manner and to provide support at the time the person needs it.

The overall aim of the E-dherence Pilot study is to evaluate the feasibility of the E-Health intervention to enhance OHT adherence in BCS. Feasibility is defined based on 1.The eHealth intervention acceptability, 2. eHealth intervention quality and 3. medication adherence.

The study will include female breast cancer starting their first prescription of tamoxifen or aromatase inhibitors and are outpatient and followed-up in either of the 2 study sites. Participants should be 18 years or older and be fluent in french and or German and possess a smart-phone (iOS, Android). The investigators exclude males, patients with in situ metastatic tumors, inpatients and non Luxembourg residents.

Within the E-dherence Pilot study each patient receives the eHealth intervention.

The eHealth intervention consists a Medication Event Monitoring Systems (MEMS®) Helping Hand and MEMS Adherence Software application.

The eHealth intervention will support BCS to adhere to the recommended OHT (i) by alerting the participants to take their OHT, and (ii) by allowing patient-physician communication.

The intervention consists of a Medication Event Monitoring Systems (MEMS®), an electronic pillbox that counts the OHT intake, the date and time. Through Near Field Communication (NFC) the device is connected to the MEMS Adherence Software application on the patients' phone (Android or iOS). At the beginning, each patient can personalize the application. This application registers the history of OHT adherence (time and date of medication intake) and sends reminders to the patient to take the treatment as scheduled.

Additionally, the patient receives an integrated calendar in the App that notifies the patient for upcoming medical visits. The eHealth intervention comprises a questionnaire that should be filled-out weekly and that informs about the presence and severity of side effects. These data are collected in real-time and monitored on a weekly basis by the clinical research nurse (CRN) in charge of the study. In case of an alert, meaning recurrent non-adherence and/or reporting of side-effects, the CRN will contact the breast cancer nurse (BCN) in charge of the patient. Thus the BCN will contact the patient by phone to check on their health status and together define the future procedure in order for the patient to remain on OHT and/or to better manage their side-effects. In a worst case scenario, the BCN will refer the patient to see the emergency department and/or the oncologist.

The study received all ethical approvals.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Female aged ≥18 years old
* 1st prescription of adjuvant treatment (Nolvadex, Arimidex)
* Treated in either the Centre Hospitalier du Luxembourg (CHL) or Centre Hospitalier Emile Mayrisch (CHEM)
* Luxembourg resident
* Fluent in French and/or German
* Outpatient
* Possession of a smart-phone (iOS, Android)

Exclusion Criteria:

* Male
* In situ or metastatic tumors
* Follow-up treatment outside of CHL or CHEM
* Non-Luxembourgish residents
* Inpatient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 3 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of medication adherence support tool | 3 months
  Proportion of patients that fully adhere to the eHealth intervention(MARS). The uMARS is a 23-item questionnaire divided into quality subscales and subjective quality. The questionnaire entails a section about the Perceived impact the eHealth application has on medication adherence.
  Medication adherence will be measured through the MEMS® Helping Hand that is connected to the MEMS Adherence Software application. Side-effects reporting are measured through a weekly questionnaire within the MEMS Adherence Software application.
Quality of medication adherence support tool | 3 months
  user Mobile Application Rating Scale (uMARS): The uMARS is a 23-item questionnaire divided into quality subscales ((a) engagement, (b) functionality, (c) aesthetics and (d) information) and subjective quality. Also, the questionnaire entails a section about the Perceived impact the eHealth application has on medication adherence. The items are scored based on a 5 point scale.
Medication Adherence | 3 months
  Proportion of days covered by medication intake during 3-months of follow-up. This outcome is measured with the Medication Event Monitoring Systems (MEMS®) Helping Hand and MEMS Adherence Software application

SECONDARY OUTCOMES:
Breast Cancer nurses phone calls to patient | 3 months
  Number of phone calls to the patients
Breast cancer nurse intervention | 3 months
  Capture of the type of intervention: Motivational; Strategic or Informational
Quality of life is measured using the EORTC Quality of Life Questionnaire (QLQ C-30) questionnaire | through study completion, an average of 3 months
  The EORTC QLQ-C30 is a health related quality of life questionnaire specific for cancer patients. It has been translated and validated into French and German. The questionnaire is divided into five functional scales, three symptom scales, one global health/ quality of life scale and a number of single items assessing additional symptoms commonly reported by cancer patients. The functional scales, symptom scales, and single items assessing additional symptom have a 4-point scale whereas the global health/ quality of life scale has a 7-point scale. A high score in the functional scale represents a healthy level of functioning. A high score in the global health/ quality of life scale represents a good quality of life. A high score for the symptom scale represents a high level of symptomatology. The EORTC QLQ-C30 is evaluated at baseline and end of study.
Beliefs about Medicine Questionnaire (BMQ) | through study completion, an average of 3 months
  The BMQ is an 18-item tool that assess the beliefs about treatment and has been translated and validated into French and German. The items are divided into specific treatment beliefs and general treatment beliefs the items have a 5 point Likert scale, ranging from 1 "strongly agree" to 5 "strongly disagree". For each, a total score was computed by adding together items' reverse scores. Each specific belief scores between 5 and 25, and each general belief between 4 and 20.Higher values represent stronger beliefs. The BMQ is evaluated at baseline and end of study.

CONTACTS AND LOCATIONS:
Locations (2):
- Luxembourg (2):
  - Centre Hospitalier Emile Mayrisch (CHEM), Esch-sur-Alzette
  - Centre Hospitalier de Luxembourg (CHL), Luxembourg

IPD SHARING:
Plan to Share IPD: No